CLINICAL TRIAL: NCT06106230
Title: Bee Venom Phonophoresis on Mild to Moderate Localized Plaque Psoriasis on Knee Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, lectrurer of physical therapy for general surgery and dermatology, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/2111/MTI.PT/2309292
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: randomize controlled trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A:Bee venom phonophoresis + Conservative care (Experimental): Bee venom phonophoresis + Conservative care (32 patients)
  Interventions: Combination Product: Bee venom phonophoresis
- Group B:Bee venom topical application + Conservative care (Experimental): Bee venom topical application + Conservative care (32 patients)
  Interventions: Combination Product: Bee venom phonophoresis
- Group C:Conservative care (Sham Comparator): Control group Conservative care only (32 patients) Plain gel instead of BV gel plus off ultrasound (sham ultrasound) with medical treatment
  Interventions: Combination Product: Bee venom phonophoresis

INTERVENTIONS:
Combination Product: Bee venom phonophoresis — Bee venom gel preparation with low freq ultrasound Bee venom solution (100 mg/mL) that was prepared and preserved at the correct temperature was purchased from the Egyptian Organization for Biological Products & Vaccines (Vacsera). The solution was a mix of a crude form of BV dissolved in sterile normal saline with a concentration ratio of 1:1 vol/vol. Then, the BV gel was prepared at the laboratories of the Faculty of Pharmacy, Modern University, Cairo, Egypt, by dissolving the previous mixture in 10% propylene glycol, followed by the addition of 0.01% butylparaben. To make bee venom gel, the resulting mixture was mixed with the matrix. The BV gel had a homogeneous and translucent appearance and a pH of 7.53. There was no discoloration, phase separation, or off-putting odor. Stratification was not observed after 30 min of centrifugation at 2,500 rpm at 25◦C, used with low frequency ultrasound Device: low intensity ultrasound
  Other Names: low intensity Ultrasound with bee venom gel

SUMMARY:
Chronic plaque psoriasis, or psoriasis vulgaris, is a chronic inflammatory skin disease characterized by well demarcated, erythematous, scaly plaques on the extensor surfaces of the body and scalp. The lesions may occasionally itch or sting, and may bleed when injured. Dystrophic nail changes or nail pitting are found in more than one third of people with chronic plaque psoriasis, and psoriatic arthropathy occurs in 1% to more than 10%. The condition waxes and wanes, with wide variations in course and severity among individuals.

DETAILED DESCRIPTION:
Apitherapy is an alternate therapy that relies on the usage of honeybee products, most importantly bee venom for the treatment of many human diseases. The venom can be introduced into the human body by manual injection or by direct bee stings. Bee venom contains several active molecules such as peptides and enzymes that have advantageous potential in treating inflammation and central nervous system diseases, such as Parkinson's disease, Alzheimer's disease, and amyotrophic lateral sclerosis. Moreover, bee venom has shown promising benefits against different types of cancer as well as anti-viral activity, even against the challenging human immunodeficiency virus (HIV). Many studies described biological activities of bee venom components and launched preclinical trials to improve the potential use of apitoxin and its constituents as the next generation of drugs.

Chronic plaque psoriasis is the most common form of psoriasis, accounting for more than 80% of cases. It is a chronic relapsing and remitting condition that presents as symmetrical, well-demarcated, erythematous thickened plaques with overlying silver scales. Appearance can vary depending on skin colour, ranging from pink on lighter skin to brown, purple, or grey on darker skin. It commonly affects the extensor surfaces (elbows and knees), scalp, trunk, and gluteal fold, but may arise on any part of the body. Plaques may coalesce to involve extensive areas of the skin, especially on the trunk and limbs.

ELIGIBILITY:
Inclusion criteria

* Symmetrical mild-to-moderate chronic plaque psoriasis
* Chronic stable plaque psoriasis
* Bilateral lesions of approximately 25 cm²
* Had not been receiving any treatment for at least one month.
* Those with infection or malignancy and/or subjects who had undergone major surgery in the past 6 months were not included in the study.
* Patients that had not undergone systemic treatment for psoriasis during the previous 3 months were included in the study
* age 20 - 50 with mild to moderate knee plaque psoriasis
* Symmetrical plaque psoriasis
* PASI score affected < 20
* BSA of knee involvement : 2% to 20%

Exclusion criteria

* Patients with malignant tumors, those diagnosed with psoriatic arthritis or any other systemic inflammatory disease, or those using medication were excluded from the study.
* Pregnancy
* Receiving steroid preparations
* topical or UVB therapy within previous 4 wks
* Systemic corticosteroids, PUVA, or laser phototherapy within previous 4 wks
* Other systemic therapies or biologicals within previous 3 wks
* Widespread psoriasis
* Hypercalcaemia
* Liver or renal disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Neutrophils / Lymphocyte Ratio (Neutrophil-to-Lymphocyte Ratio) | base line after 12 weeks
  Ratio
C-reactive protein (CRP) | base line after 12 weeks
  A C-reactive protein (CRP) test measures the level of C-reactive protein in your blood.
(ESR) erythrocyte sedimentation rate | base line after 12 weeks
  ESR

SECONDARY OUTCOMES:
PASI score | base line after 12 weeks
  Psoriasis area severity index (PASI), which evaluates the degree of erythema, induration, and desquamation in the affected body areas, is one of the most commonly used scales to classify disease severity
Isokinetic machine proprioceptive test | base line after 12 weeks
  A dynamometer (System 3 Pro; Biodex Medical Inc., Shirley, NY, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Ahmed Abdelhady, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Evaluation of Knee Proprioception and Factors Related to Parkinson's Disease — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5031852/
- See also: Quantitative Assessment of Proprioception Using Dynamometer in Incomplete Spinal Cord Injury Patients: A Preliminary Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5426262/